CLINICAL TRIAL: NCT00006260
Title: A Phase II Study Of An OutPatient Three Day VIP Regimen With Oral Mesna For Metastatic Breast Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Scot C. Remick, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU4196; P30CA043703 (NIH); CWRU-4196; BMS-CRWU-4196; NCI-G00-1854
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cisplatin; Etoposide; Ifosfamide; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cisplatin — cisplatin IV over 30 minutes on days 1-3.
Drug: etoposide — etoposide IV over 60-90 minutes on days 1-3.
Drug: ifosfamide — ifosfamide IV over 30 minutes on days 1-3.
Drug: Mesna — Mesna is administered IV over 15 minutes 30 minutes prior to and 4 hours after ifosfamide, then orally at 8 hours post infusion.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Drugs such as mesna may be effective in preventing some of the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy consisting of etoposide and ifosfamide given with mesna, and cisplatin in treating patients who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate in patients with metastatic breast cancer treated with etoposide, ifosfamide with mesna, and cisplatin.
* Determine the tolerability and toxicity of this regimen in these patients.

OUTLINE: Patients are stratified according to number of prior chemotherapy courses for metastatic disease (0 vs 1).

Patients receive etoposide IV over 60-90 minutes, cisplatin IV over 30 minutes, and ifosfamide IV over 30 minutes on days 1-3. Mesna is administered IV over 15 minutes 30 minutes prior to and 4 hours after ifosfamide, then orally at 8 hours post infusion. Treatment continues every 28 days in the absence of unacceptable toxicity or disease progression.

Patients are followed every 3 months.

PROJECTED ACCRUAL: At least 36 patients (16 per stratum) will be accrued over 36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven progressive metastatic breast cancer
* Measurable disease

  * Any lesion measurable in 2 dimensions
  * Hepatic metastases if the sum of the measurements below the costal margin in the midclavicular line and the tip to the xiphoid process is greater than 5 cm during quiet respiration
  * Hepatic defects that are clearly measurable by radionuclide, CAT, or MRI scans
  * Bone metastases are not considered measurable disease
  * Evaluable disease allowed if measurable disease also present
* No brain metastases, carcinomatous meningitis, or spinal cord compression
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* Not specified

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Hemoglobin at least 10 g/dL
* WBC at least 4,000/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL

Renal:

* Creatinine no greater than 1.5 mg/dL
* No bladder outlet obstruction

Cardiovascular:

* No symptomatic cardiovascular disease (e.g., congestive heart disease) or inability to tolerate a fluid load

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection
* No prior malignancies except adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No greater than 1 prior biologic response modifier treatment for metastatic disease

Chemotherapy:

* No greater than 1 prior chemotherapy regimen for metastatic disease allowed
* Patients who relapsed during or within 6 months after adjuvant chemotherapy are considered to have failed 1 regimen
* Patients who relapsed more than 6 months after adjuvant chemotherapy are considered to not have had a prior regimen
* Greater than 4 weeks since prior chemotherapy (greater than 6 weeks for mitomycin or nitrosoureas) and recovered
* No prior cisplatin, etoposide, or ifosfamide

Endocrine therapy:

* Prior medical or surgical hormonal therapy allowed

Radiotherapy:

* Prior radiation therapy to areas of measurable disease allowed if indicator lesion increased in size by greater than 25% after treatment
* Recovered from effects of prior radiotherapy

Surgery:

* Recovered from effects of major surgery

Other:

* At least 7 days since prior nephrotoxic drugs (e.g., aminoglycosides, diuretics, lithium, intravenous contrast, or nonsteroidal antiinflammatory drugs)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 1997-05; Primary Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Determine the objective response rate in patients with metastatic breast cancer treated with etoposide, ifosfamide with mesna, and cisplatin. | Treatment continues every 28 days in the absence of unacceptable toxicity or disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Scot C. Remick, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Viana LV, Leitao CB, Grillo MF, Rocha EP, Brenner JK, Friedman R, Gross JL. Hypertension management algorithm for type 2 diabetic patients applied in primary care. Diabetol Metab Syndr. 2013 Sep 12;5(1):52. doi: 10.1186/1758-5996-5-52. PMID 24028306